CLINICAL TRIAL: NCT01567514
Title: A 2-year Clinical Study on Postoperative Pulpal Complications Arising From the Absence of a Glass-ionomer Lining in Deep Occlusal Resin Composite Restorations
Brief Title: Postoperative Pulpal Complications in Posterior Resin Composite Restorations Without Glass-ionomer Cement Lining
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-IRB 2008/269.3110
Record Dates: First submitted 2012-03-28; First posted 2012-03-30 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Dental Caries
Keywords: Deep occlusal caries restored with resin composite; on Pit and Fissure Surface Penetrating Into Dentin
MeSH Terms: conditions — Dental Caries | interventions — Fuji glass-ionomer lining cement; Vitrabond

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glass-ionomer cement lining (Active Comparator): Presence of glass-ionomer cement lining in posterior resin composite restorations.
  Interventions: Procedure: Glass ionomer cement lining
- No glass-ionomer cement lining (No Intervention): Absence of glass-ionomer cement lining in posterior resin composite restorations
  Interventions: Procedure: Glass ionomer cement lining

INTERVENTIONS:
Procedure: Glass ionomer cement lining — Resin-modified glass ionomer lining
  Other Names: Vitrebond (3M ESPE, St. Paul, MN, USA)

SUMMARY:
The purpose of this study is to observe the effects of glass-ionomer cement (GIC) lining on risk of pulpal complications in deep occlusal cavities with resin-based restorations.

DETAILED DESCRIPTION:
Fifty three patients aged 18-30 years who had one or two deep occlusal carious lesions (≥ 3 mm in depth) in molars were recruited. Dental caries was removed and the prepared cavity was restored with resin composite using one of two restorative procedures: (1) without GIC lining; (2) with (resin-modified) GIC lining. Restored teeth were evaluated for any pulpal complications (subjective symptoms, objective signs or loss of tooth vitality) at one month (baseline), one year and two years after restoration.

ELIGIBILITY:
Inclusion Criteria:

* Deep dental caries on occlusal surfaces of molar teeth

Exclusion Criteria:

* Shallow and moderate-depth caries
* Caries exposed pulp

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Postoperative pulpal complications | 2 years
  Signs and symptoms (subjective/objective) of pulpal & periapical diseases. Response to electrical pulp testing.

CONTACTS AND LOCATIONS:
Overall Officials: Emeritus Prof. Harold Messer, Ph.D., Study Director — University of Melbourne
Locations (1):
- Faculty of Dentistry, Mahidol University, Bangkok, Thailand